CLINICAL TRIAL: NCT02085759
Title: Th2 Cytokine Responses in Overweight/Obese Subjects
Brief Title: T-helper 2 (Th2) Cytokine Responses in Overweight/Obese Subjects
Status: Completed | Type: Observational
Sponsor: West Penn Allegheny Health System (Other)
Collaborators: Pennsylvania Allergy and Asthma Research Foundation (Unknown)
Responsible Party: Principal Investigator, David Skoner, MD, Director, Allergy and Asthma Institute, West Penn Allegheny Health System
Other Study IDs: RC# 4729
Record Dates: First submitted 2009-05-28; First posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Overweight; Obesity
Keywords: Healthy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal BMI: Subjects with a BMI range of 18.5 to 24.9 which is defined by the CDC as within normal range.
- Overweight BMI: Subjects with a BMI of 25.0 to 29.9 are defined by the CDC as being overweight.
- Obese BMI: Subjects with a BMI of 30.0 and above are defined by the CDC as being obese.

SUMMARY:
Cytokines are chemicals that are naturally made by your body. Certain cytokine levels are changed in the blood of patients who develop allergies and/or asthma. Cytokine levels may also be changed in some individuals who are overweight or obese. The purpose of this study is to determine if certain cytokine levels differ based on a person's weight and whether or not they have allergies or asthma. Information gathered in this study will be compared to information gathered from subjects who have participated in another similar study for patients who have allergies and/or asthma.

DETAILED DESCRIPTION:
The aims of this study are to:

1. Characterize the relationship between BMI and Th2 skewing in non-atopic adult subjects.
2. Compare these results to those previously obtained from atopic adult subjects It is expected that the results of this study will demonstrate enhanced Th2 skewing in overweight and obese atopic subjects as compared to non-atopic subjects. It is further anticipated that the results of this study will be used as preliminary data to generate an NIH grant application exploring the link between obesity and atopy.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 to 50 years
* pre-bronchodilator FEV1 > 80% predicted with no evidence of reversibility following administration of bronchodilator
* no history of allergies

Exclusion Criteria:

* medical history consistent with atopy and/or asthma
* any positive response to allergy skin testing for inhalant allergens (defined as a wheal > 3 mm larger than the negative control)
* a pre-bronchodilator FEV1 < 80% predicted
* > 12% reversibility in FEV1 following administration of a bronchodilator
* any history of significant chronic illness
* history of respiratory infection within the past 2 weeks
* any use of prescription medications other than oral contraceptives or thyroid hormone replacement within the past 2 months
* use of any investigational medication within the past month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be male or female, aged 18-50 years, and of any race. Subjects must be healthy with no history of allergies or asthma. Subjects will be placed in one of three groups based on their BMI: normal, overweight, or obese.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Th2 Cytokine levels | Baseline (only visit)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoner, MD, Principal Investigator — Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute); Deborah Gentile, MD, Study Director — Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Locations (1):
- Allegheny General Hospital, Dept. of Allergy, Asthma, & Immunology, Pittsburgh, Pennsylvania, United States